CLINICAL TRIAL: NCT01479257
Title: Determinants of Multiple Health Risk Behaviors Among Latinos
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2011-0696; 1K01CA157689 (NIH); R25T CA57730 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Risk Factors in Latinos
Keywords: Cancer; Risk factors; Latinos; Hispanic Americans; Hispanics; Latino resident; Houston metropolitan area; Spanish speaking; Cancer risk behaviors; Questionnaires; Surveys; Accelerometer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bilingual Latinos: Bilingual Houston area Latinos surveyed for 7 continuous days with objective and subjective assessments using accelerometer and smart phone.
  Interventions: Behavioral: Questionnaires; Device: Accelerometer; Device: Smart Phone

INTERVENTIONS:
Behavioral: Questionnaires — 36 questionnaires at the first visit (a total of 474 questions) and 25 questionnaires at the second visit (a total of 278 questions), taking about 60 to 90 minutes to complete each visit.
  Other Names: Surveys
Device: Accelerometer — Small device worn on the hip for 7 consecutive days that measures physical activity.
  Other Names: Movement meter
Device: Smart Phone — Questions on smart phone up to 5 times a day for 7 days taking about 5-7 minutes to complete each time.
  Other Names: cell phone

SUMMARY:
The goal of this research study is to learn how cultural, environmental, and interpersonal experiences, as well as personal thoughts and feelings, influence cancer risk behaviors among Latino residents of Houston, Texas.

DETAILED DESCRIPTION:
Study Participation:

If you are eligible and choose to take part in this study, you can choose to visit the clinic 2 times or have research staff visit you in your home or a community setting (such as a church or community center) 2 times.

At the first visit (this is the same visit where you complete the in-person screening test):

* You will have your height, weight, and waistline measured.
* You will be given a smart phone to take home with you. You will answer questions on the smart phone up to 5 times a day for 7 days. The phone will beep at random times (4 times per day) and set times (in the evening) to prompt you to answer questions about what you are doing and your current thoughts and feelings. These questions should take about 5-7 minutes to complete each time.
* You will be given an accelerometer (a movement meter). The accelerometer is a small device worn on your hip that measures the amount of physical activity you do. You will wear the accelerometer for 7 days in a row.
* You will receive training on how to use the smart phone and the accelerometer.

At the second visit, you will return the smart phone and the accelerometer.

At both study visits, you will be asked to complete questionnaires that ask about your feelings, moods, and behaviors. You will complete 36 questionnaires at the first visit (a total of 474 questions) and 25 questionnaires at the second visit (a total of 278 questions). These questionnaires should take about 60 to 90 minutes to complete.

Throughout the study, you will be contacted by mail, email, or telephone for reminders of visits. You will be reminded before each visit. You will be asked to provide the names and contact information for family and/or friends should the study staff have trouble reaching you.

Confidentiality:

Each time you complete a survey on the smart phone, your answers will be saved on the phone. When you return the phone, all of your answers will be downloaded from the phone to a secure server, where they will be stored. Then, all of your information will be deleted from the phone. Your name or other personal information will not be stored on the phone.

Your name and other identifying information will not be stored together in the same files as other information you provide during your participation in the study. The link between your identifying information and other data will be kept in a separate file and securely protected. The link between you and the study data will be destroyed 5 years after the study ends.

Length of Study:

You will be considered off study when you complete the second visit.

This is an investigational study.

Up to 225 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as Latino in ethnicity
2. Are between the ages of 18-65, inclusive
3. Possess a valid home address and functioning telephone number
4. Possess marginal to adequate health literacy in English (as indicated by a score of at least 45 on the Rapid Estimate of Adult Literacy in Medicine) and Spanish (as indicated by a score of at least 38 on the Short Assessment of Health Literacy for Spanish Adults).

Exclusion Criteria:

1. Used an illicit substance in the past 30 days
2. Another household member enrolled in the study
3. Pregnant or breastfeeding
4. Participated in a smoking cessation program in the last 90 days
5. Uses nicotine replacement products
6. Uses other tobacco products besides cigarettes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bilingual Latinos in the Houston, Texas metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Determinants of Cancer Risk Behaviors in Latinos | 7 days
  Outcomes assessed through daily diary ecological momentary assessment (EMA) data and coded as yes (engaged in activity) or no (did not engage in activity). EMA assessments done over 7 contiguous days in a questionnaire computer-administered self-interview format.

CONTACTS AND LOCATIONS:
Overall Officials: Larkin L. Strong, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org